CLINICAL TRIAL: NCT00849433
Title: Effects of Smoking on Airway Remodeling and Phenotypic Changes of the Airway Epithelium in Asthma and COPD: Strategies to Restore the Epithelial Barrier, Repair and Steroid Sensitivity.
Brief Title: Effects of Smoking on Bronchial Epithelium
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, doctor, University Medical Center Groningen
Other Study IDs: METc2009008
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Asthma; Copd
Keywords: Inflammation; epithelial; integrity; ECIS
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchial biopsies Bronchial brushes Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 30 patients with asthma
- 2: 30 patients with COPD

SUMMARY:
Asthma and chronic obstructive pulmonary disease (COPD) are chronic inflammatory airway diseases affecting millions of people worldwide. Inhaled corticosteroids (ICS) are by far the most effective treatment with a broad anti-inflammatory spectrum. Nevertheless, most COPD patients and a proportion of severe asthma patients are corticosteroid-resistant (CR) and to fail to respond to ICS even when higher doses are given. These corticosteroid-resistant patients suffer from persistent symptoms and repeated asthma exacerbations. It has been suggested that smoking and oxidative stress may induce corticosteroid-resistance. The reactive oxygen species (ROS) responsible for oxidative stress can be generated exogenously (air pollutants, cigarette smoke) and endogenously by metabolic reactions. After inhaling air pollutants or cigarette smoke, the bronchial epithelium is exposed. Preliminary data from our own lab suggest that smoking and oxidative stress may decrease epithelial cell-cell contact formation. This results not only in a decreased barrier function, but also in an increased production of pro-inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with allergic asthma:

* Age between 18 and 65 years.
* < 10 packyears, no smoking in the last year.
* The presence of allergy defined as at least one positive wheal/flare reaction (2 mm relative to control) to a skin prick test with sixteen common aero-allergens).
* FEV1 > 80% predicted.
* PC20 methacholine or PC20 histamine < 8 mg/ml.

Inclusion criteria for patients with COPD:

* Age between 45-75 years.
* ≥ 10 packyears.
* FEV1 between 30% and 80% of predicted.

Exclusion criteria:

* Any disease that, as judged by the Investigator, could have affected the outcome of this study.
* A respiratory tract infection within 4 weeks of the start of the study.
* A history of life-threatening asthma, defined as exacerbation of asthma or COPD that required intubation or was associated with hypercapnea.
* History of myocardial infarction or documented myocardial ischemia.
* Pregnancy, or the possibility of being pregnant (a pregnancy test will be performed in women of childbearing potential who do not use adequate anticonception as judged by the investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with asthma; 30 patients with COPD
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Epithelial integrity as measured with ECIS | 2 years

SECONDARY OUTCOMES:
Inflammatory cells and mediators | 2 years
Production of inflammatory cytokines | 2 years
Markers of epithelial integrity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, MD, PhD, Principal Investigator — University Medical Center Groningen; Dirkje S Postma, Professor, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands